CLINICAL TRIAL: NCT03690492
Title: The Box 2.0: Using Smart Technology for Early Diagnosis of Complications After Cardiovascular Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, RoderickTreskes, Principal Investigator, Leiden University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NL65959.058.18
Record Dates: First submitted 2018-09-24; First posted 2018-10-01 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Rehabilitation After Cardiovascular Surgery; Mobile Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The Box 2.0 (Experimental): Patients will be given a Box, in which they will find a thermometer, blood pressure monitor, activity tracker, weight scale, blood oxygen saturation monitor, a single lead ECG device and a four lead ECG device. Also, they will be followed-up by use of two webcam consultations instead of a normal outpatient clinic visit.
  Interventions: Other: The Box 2.0
- Controls (No Intervention): Patients will not receive a Box. They will be followed up by standard care, returning to the outpatient clinic at the same frequency and timing as The Box 2.0 arm.

INTERVENTIONS:
Other: The Box 2.0 — Patients in the intervention arm will receive a Box with several devices that is hypothesized to allow for better and earlier detection of complications after cardiac surgery.
  Arms: The Box 2.0

SUMMARY:
The objective of this study is to determine the effect on quality of care when introducing smart technology in patients who underwent cardiovascular surgery. Patients who consent to take part in the study, receive a box containing two smartphone compatible ECG monitors, an oxygen saturation monitor, a weight scale, a thermometer, an activity tracker and a blood pressure monitor. They will be followed up by replacing one of the outpatient clinic visits by an e-consult, in which a patients does not have to go to the hospital. Instead, he or she will talk with his or her doctor or nurse practitioner via a secured video connection. The primary endpoint of the study will be the diagnosis of atrial fibrillation within 3 months after cardiac surgery.

DETAILED DESCRIPTION:
Over the past five years, smartphone compatible detectors of cardiovascular disease parameters have been released on the consumers market. Examples of these include heart rate monitors, ECG monitors, blood pressure monitors, activity trackers and fat percentages monitors. These monitors have often been validated and are CE-marked for use in the European Union within their intended use.

Recent publications implicate that home monitoring with such consumer devices might improve quality of care. A study by Bosworth et al. in patients with hypertension showed that increased monitoring and subsequent treatment led to a better controlled blood pressure in patients who were treated for hypertension. Another study, which is currently being carried out at the LUMC, is investigating whether patients benefit from a smart technology intervention after they had a myocardial infarction. Preliminary (unpublished) results show that clinical outcomes are similar, with higher patient satisfaction. Cost analyses show that there is a cost reduction per patient with smart technology follow-up. Therefore, smart technology could be a useful tool to improve patient monitoring and therefore patient safety.

Patients who are discharged after they underwent cardiovascular surgery are at risk to develop one or more of three most seen late complications: sternal wound infection, cardiac decompensation or rhythm disturbances such as atrial fibrillation. This is not always detected before those patients are discharged.

Currently, patients who underwent cardiovascular surgery return to the outpatient clinic 14 days and three months after discharge. They are seen by a specialist nurse or cardiologist, who will perform a general check-up and inspect the sternal wound. An echocardiogram will be performed before the three-month visit. If there is suspicion for a rhythm disturbance on the outpatient clinic visit, the cardiologist might decide to perform Holter monitoring during 24 hours. As this is a small window of time, not all rhythm disturbances will be diagnosed. Smart technology is hypothesized to increase the chances of diagnosing rhythm disturbances. In the case of sternal wound infection and cardiac decompensation, smart technology may show a declining trend before a patient visits the outpatient clinic, which can lead to early detection and treatment.

A small pilot study by McElroy et all found that after cardiovascular surgery, both the patient as well as the health care team are highly satisfied with added smart technology, due to the ease of use of the technology and platform. There was a main focus on readmission rates, which did not differ between the groups. However the trend shows an increase in diagnosing atrial fibrillation (15,4 vs 29,6%), sternal wound infection or cardiac decompensation were not studied.

To our knowledge, no other study has yet looked into diagnosing late complications after cardiovascular surgery with the help of smart technology. It is hypothesized that smart technology could help diagnose the main three diagnoses mentioned above early on and with that, improve quality of care in patients after cardiovascular surgery. Therefore, in this study, the clinical effectiveness of a smart technology intervention is investigated in patients who have underwent cardiovascular surgery at the department of Thoracic Surgery at Leiden University Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoes cardiovascular surgery: CABG, valve reconstruction or replacement, aortic root or ascending aortic surgery, or any other cardiothoracic surgery performed by median sternotomy such as atrial or ventricular septal defect closure, Dor or Morrow procedure, cardiac tumor removal and/or surgical treatment of coronary artery anomalies.
* Patient is able to communicate in English or Dutch
* Patient has been referred by a cardiologist from the Leiden University Medical Center, Cardiological Center Voorschoten, Alrijne Hospital or Haaglanden Medical Center

Exclusion Criteria:

* Patient is < 18 years old
* Patient is pregnant
* Patient is considered an incapacitated adult
* Patient is unwilling to sign the informed consent form
* Patient undergoes emergency thoracic surgery (INTERMACS 1 or 2)
* Patient has active endocarditis at the time of operation
* Patient is on mechanical circulatory support before operation
* Patient has a ventricular septal rupture
* Patient undergoes extracorporeal membrane oxygenation or ventricular assist device insertion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Dectection of and time to detection of atrial fibrillation | Until 3 months after surgery
  Diagnosis of atrial fibrillation and the time it took a subject to reach that outcome, measured in both study arms

SECONDARY OUTCOMES:
Dectection of and time to detection of cardiac decompensation | Until 3 months after surgery
  Diagnosis of cardiac decompensation and the time it took a subject to reach that outcome, measured in both study arms
Quality of Life (QoL) | 3 months after surgery
  QoL of both study arms, using the EQ-5D-5L (Dutch translation)
Patient satisfaction of care | 3 months after surgery
  Satisfaction in both study arms, using a modified PSQ-18 (Dutch translation)
Overall mortality | 3 months after surgery
  Mortality in both study arms
Major adverse cardiac events | Until 3 months after surgery
  Either cardiac death, myocardial infarction, cardiac tamponade, TIA or ischaemic stroke
Re-admission to either the cardiology or thoracic surgery ward | Until 3 months after surgery
  Re-admission in both study arms
Total amount of cardiology related visits to an emergency department until three months after discharge | Until 3 months after surgery
  ER visits (at the Leids University Medical Center, Alrijne Ziekenhuis or Haaglanden Medisch Centrum) in both arms
Blood pressure control | 3 months after surgery
  BP control in both study arms, both systolic and diastolic
Cost-effectiveness | 2 years
  Cost-effectiveness of the intervention
Detection of and time to detection of sternal wound infection | Until 3 months after surgery
  Diagnosis of sternal wound infection and the time it took a subject to reach that outcome, measured in both study arms

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Centre, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Biersteker TE, Boogers MJ, de Lind van Wijngaarden RA, Groenwold RH, Trines SA, van Alem AP, Kirchhof CJ, van Hof N, Klautz RJ, Schalij MJ, Treskes RW. Use of Smart Technology for the Early Diagnosis of Complications After Cardiac Surgery: The Box 2.0 Study Protocol. JMIR Res Protoc. 2020 Apr 21;9(4):e16326. doi: 10.2196/16326. PMID 32314974